CLINICAL TRIAL: NCT03391232
Title: Safety, Tolerability, Immunogenicity and Efficacy of Multiple PolyPEPI1018 Vaccinations as an Add-on Immunotherapy to the Standard-of-Care Maintenance Therapy in Subjects With Metastatic Colorectal Cancer
Brief Title: PolyPEPI1018 Vaccine and CDx for the Treatment of Metastatic Colorectal Cancer (OBERTO)
Acronym: OBERTO
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Treos Bio Zrt (Industry)
Collaborators: Mayo Clinic (Other); University of Pisa (Other); Laboratory Corporation of America (Industry); PPD Development, LP (Industry); ImmunXperts SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OBERTO 101
Record Dates: First submitted 2017-12-19; First posted 2018-01-05 (Actual); Results first posted 2022-04-14 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PolyPEPI1018 CRC Vaccine (Experimental): The vaccine contains 6 synthetic peptides mixed with the adjuvant Montanide™. The peptides were selected to induce T cell responses against 12 dominant epitopes from 7 cancer testis antigens (CTAs), which are the most frequently expressed CTAs in colorectal cancer. The 6 peptides were optimized to induce long lasting CRC specific T cell responses.
  Interventions: Biological: PolyPEPI1018 CRC Vaccine

INTERVENTIONS:
Biological: PolyPEPI1018 CRC Vaccine — Colorectal Cancer Vaccine

SUMMARY:
Phase I/II clinical trial investigates the safety, tolerability, immunogenicity and preliminary efficacy of multiple doses of PolyPEPI1018 CRC vaccine as an add-on treatment to the standard-of-care maintenance therapy in patients with metastatic colorectal cancer. Clinical responses will be evaluated by indiction of T cell responses, T lymphocyte infiltration in accessible biopsy sites, and by objective tumor responses. This study will also explore the accuracy of the predicted T cell responses in each patient using the candidate companion diagnostic test and the correlations between clinical responses and predicted T cell responses.

DETAILED DESCRIPTION:
This is a Phase I/II, open-label, single-arm, multicenter study to evaluate the safety, tolerability, immunogenicity and efficacy of a multiple subcutaneous injection of PolyPEPI1018 as an add-on immunotherapy to the standard-of-care maintenance therapy in approximately 15 subjects with metastatic colorectal cancer.

The first part of the study investigates the administration of a single vaccine dose during 12-week follow-up period on an outpatient basis. Screening is performed in parallel with the subject's completion of the standard-of-care first-line treatment and initiation of the standard-of-care maintenance treatment. A single dose of PolyPEPI1018 is administered after the subject initiates the maintenance regimen, and within 3 weeks after the eligibility CT scan was performed. Subjects are monitored every 3 weeks for 12 weeks.

The second part of the study investigates the administration of 3 vaccine doses (Weeks 0, 13, 26) then 12 weeks follow-up on an outpatient basis.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects, 18-75 years of age at time of Screening who provide written informed consent prior to initiation of any study procedure
2. Histologically confirmed metastatic adenocarcinoma originating from the colon or the rectum
3. Presence of at least 1 measurable reference lesion according to the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 criteria
4. Experienced PR or stable disease during first-line treatment with a systemic chemotherapy regimen and 1 biological therapy regimen
5. Maintenance therapy with a fluoropyrimidine (5-fluorouracil or capecitabine) plus the same biologic agent (bevacizumab, cetuximab or panitumumab) used during induction, scheduled to initiate prior to the first day of treatment with the study drug
6. No more than 1 line of chemotherapy regimen for mCRC (adjuvant therapy for non-metastasized disease is allowed if terminated more than 6 months before Screening and without recurrence within 6 months after the end of adjuvant treatment)
7. Last CT scan at 3 weeks or less before the first day of treatment
8. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
9. Women of childbearing potential must agree to appropriately use an effective form of contraception (failure rate of <1% per year) for 3 months from the day of the treatment. An effective form of contraception is defined as using hormonal contraceptives or an intrauterine device combined with at least 1 of the following forms of contraception: a diaphragm, cervical cap or condom
10. Men must agree to use an effective form of contraception (as defined above), and not donate sperm for 3 months from the day of the treatment
11. White blood cell count ≥3.0 × 109/L with neutrophils ≥1.5 × 109/L
12. Platelets ≥100 × 109/L, hemoglobin ≥5.6 mmol/L (corresponding to 9 g/dL)
13. Serum bilirubin ≤1.5 × upper limit of normal (ULN) set by the site
14. Alanine amino transferase (ALAT) and aspartate amino transferase (ASAT) ≤2.5 × ULN in the absence of liver metastases. ALAT and ASAT ≤5 × ULN set by the site in the presence of liver metastases
15. Serum creatinine ≤1.5 × ULN set by the site and creatinine clearance >30 mL/min using Cockroft formula
16. Relevant toxicities of prior therapies must have resolved, except for oxaliplatin-related neuropathy or alopecia
17. Anticipated life expectancy ≥6 months Subject is willing and able to comply with the requirements of the protocol

Exclusion Criteria:

1. Received chronic systemic immune therapy or immunosuppressant medication other than steroids within the last 6 weeks prior to start of study treatment
2. Received continuous systemic steroid treatment within the last 2 weeks prior to start of study treatment
3. Colorectal cancer with documented high microsatellite instability (MSI-H)
4. Colorectal cancer with documented BRAF mutations
5. Pre-existing systemic autoimmune or antibody-mediated diseases or immune deficiency diseases
6. Central nervous system (CNS) metastases
7. Active or uncontrolled severe infections or undiagnosed febrile condition >38ºC
8. Acute or subacute intestinal obstruction or history of chronic intestinal inflammatory diseases
9. Symptomatic peritoneal carcinomatosis
10. Peritonitis
11. Serious, non-healing wounds, ulcers or bone fractures
12. Nephrotic syndrome
13. Arterial thromboembolisms or severe hemorrhages within 6 months before study enrolment (except bleeding tumor before tumor resection surgery)
14. Hemorrhagic diathesis or thrombotic tendency
15. Major surgery or radiotherapy within 12 weeks prior to the study treatment or anticipation of needing such procedure during the study period
16. Uncontrolled pleural effusion, pericardial effusion or ascites requiring repeated drainage more than once every 28 days
17. Participants with active malignancy (other than colorectal cancer) or a prior malignancy within the past 12 months
18. Participant with myocardial infarction within 6 months prior to enrollment or New York Heart Association Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to the first dose of study treatment, any electrocardiogram (ECG) abnormality at Screening must be documented by the investigator as not medically relevant
19. Administration of a live, attenuated vaccine within 4 weeks before randomization or anticipation of a live attenuated vaccine will be required during the study
20. Participant has participated in another clinical study involving an investigational product (IP) or investigational device within 30 days prior to enrollment or is scheduled to participate in another clinical study involving an IP or investigational device during the course of this study
21. Known hypersensitivity to any component of the investigational drug
22. If female, participant is pregnant (exclusion confirmed with beta-human chorionic gonadotropin [hCG] test) or lactating at the time of enrollment, or has plans to become pregnant or start breastfeeding during the study
23. Pre-existing alcohol or drug abuse
24. Medical or mental impairments which make it impossible to obtain the patient's consent or to conduct the study
25. A significant concomitant medical condition which the clinical investigator believes precludes the patient from enrolling in the study Absent or limited legal competence

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-05-03 (Actual); Primary Completion 2019-07-17 (Actual); Study Completion 2019-07-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eva Vegh, MD, MDA, Study Chair — Treos Bio Zrt
Locations (2):
- Mayo Clinic, Rochester, Minnesota, United States
- Universiti di Pisa, Pisa, PI, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hubbard JM, Toke ER, Moretto R, Graham RP, Youssoufian H, Lorincz O, Molnar L, Csiszovszki Z, Mitchell JL, Wessling J, Toth J, Cremolini C. Safety and Activity of PolyPEPI1018 Combined with Maintenance Therapy in Metastatic Colorectal Cancer: an Open-Label, Multicenter, Phase Ib Study. Clin Cancer Res. 2022 Jul 1;28(13):2818-2829. doi: 10.1158/1078-0432.CCR-22-0112. PMID 35472243
- See also: Treos Bio uses novel biomarkers to develop personalized and off-the-shelf cancer vaccines — http://www.treosbio.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The participants were recruited based on physicians referral at two medical centers between May and Dec 2018. The first subject was enrolled on 3 May 2018 and the last subject was enrolled on 13 Dec 2018.
Pre-assignment Details: Of 13 screened participants 11 met the inclusion criteria and were enrolled and treated. One of the two not enrolled subjects were over 75 years (IN01), and the other had the last CT scan over 3 weeks (IN07). All 11 subjects started and completed Part A to get the first dose and 6 of them continued treatment in Part B for additional doses (Amended protocol).
Groups:
- Single Dose - PolyPEPI1018 CRC Vaccine: The subjects in this group received only one dose of PolyPEPI1018 CRC vaccine and they finished the trial after 12 weeks follow up.
  The PolyPEPI1018 CRC vaccine contains 6 synthetic peptides derived from 7 tumor specific antigens (AG), mixed with the adjuvant Montanide™.
- Multiple Doses - PolyPEPI1018 CRC Vaccine: The subjects received 3 doses of the PolyPEPI1018 CRC vaccine Q12W. The PolyPEPI1018 CRC vaccine contains 6 synthetic peptides derived from 7 tumor specific antigens (AG), mixed with the adjuvant Montanide™.
Period: Part A - First Dose (1-12weeks)
Arm/Group | Single Dose - PolyPEPI1018 CRC Vaccine | Multiple Doses - PolyPEPI1018 CRC Vaccine
Started | 5 | 6
Completed | 5 (This cohort finished the trial here after 12 weeks.) | 6 (After interim analysis this cohort continued the trial.)
Not Completed | 0 | 0
Period: Part B - Additional 2 Doses (13-38weeks)
Arm/Group | Single Dose - PolyPEPI1018 CRC Vaccine | Multiple Doses - PolyPEPI1018 CRC Vaccine
Started | 0 | 6
Completed | 0 | 3
Not Completed | 0 | 3
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Population: All 11 subjects, Full analysis dataset
Groups:
- Single Dose of PolyPEPI1018 CRC Vaccine: The subjects were treated with only one dose PolyPEPI1018 CRC vaccine.
- Multiple Dose of PolyPEPI1018 CRC Vaccine: The subjects received 2 or 3 doses PolyPEPI1018 CRC vaccine.
- Total: Total of all reporting groups
Arm/Group | Single Dose of PolyPEPI1018 CRC Vaccine | Multiple Dose of PolyPEPI1018 CRC Vaccine | Total
Number analyzed (Participants) | 5 | 6 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.8 (5.3) | 47.5 (6.0) | 55.4 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 4 | 6 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 6 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 6 | 7
  Italy | 4 | 0 | 4
Weight [Mean (Standard Deviation); unit: Kg] | 82.6 (13.2) | 95.7 (24.9) | 89.7 (20.6)
Height [Mean (Standard Deviation); unit: cm] | 160.0 (33.7) | 185.9 (9.6) | 174.1 (26.2)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Related Adverse Events
Description: Occurrence of at least 1 ≥Grade 4 local adverse event (AE) or 1 ≥Grade 3 systemic AE and/or signs/symptoms, lab toxicities, and/or clinical events that is probably or definitely related to study treatment
Time Frame: from 1st vaccination to 21 days after last vaccinations, up to 41 weeks
Population: All subjects
Measure: Count of Participants; unit: Participants
Arm/Group | Single Dose of PolyPEPI1018 CRC Vaccine | Multiple Dose of PolyPEPI1018 CRC Vaccine
Number analyzed (Participants) | 5 | 6
Participants | 0 | 0

2. Secondary Outcome: Number of Participants Having T Cell Immune Response
Description: Measured CD4+ and CD8+ T cell responses from each subject for each antigen of the vaccine
Time Frame: 12 weeks
Population: Ten of 11 subject had sufficient PBMC samples to evaluate T cell responses
Measure: Count of Participants; unit: Participants
Arm/Group | Single Dose of PolyPEPI1018 CRC Vaccine | Multiple Dose of PolyPEPI1018 CRC Vaccine
Number analyzed (Participants) | 4 | 6
Participants
  CD4+ T cell responses | 4 | 6
  CD8+ T cell responses | 4 | 5
  CD8+ T cell responses against 3 or more AG | 4 | 4
  Booth CD4+ and CD8+ T cell responses | 4 | 5

3. Secondary Outcome: Number of Predicted Antigen Specific T Cell Responses Per Patient
Description: Epitopes restricted to multiple HLA class I alleles (Personal Epitope, PEPI) of a subject were predicted. PEPIs determined for each vaccine antigen can predict the antigen-specific T cell responses for each patient.
Time Frame: 21 days
Population: All subjects
Measure: Mean (Standard Deviation); unit: predicted PEPIs
Arm/Group | Single Dose of PolyPEPI1018 CRC Vaccine | Multiple Dose of PolyPEPI1018 CRC Vaccine
Number analyzed (Participants) | 5 | 6
predicted PEPIs | 4.80 (1.64) | 4.17 (1.33)

4. Other Pre Specified Outcome: Number of Participants With Objective Tumor Responses - Objective Response Rate (RECIST v1.1)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
  CT scans were performed at screening and weeks 6,12 after each vaccination. The objective response were based on for each subject's last CT scan evaluation.
Time Frame: 12 weeks
Population: Full set
Measure: Count of Participants; unit: Participants
Arm/Group | Single Dose of PolyPEPI1018 CRC Vaccine | Multiple Dose of PolyPEPI1018 CRC Vaccine
Number analyzed (Participants) | 5 | 6
Participants | 1 | 2

5. Other Pre Specified Outcome: Number of Participants With Objective Tumor Responses - Disease Control Rate (Best Overall Response is Partial Response or Stable Disease)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease (SD) <30% increase compare to smallest sum of the longest diameter of target lesions.
  CT scans were performed at screening and weeks 6,12 after each vaccination. The DCR were counted as the best response (PR or SD) for each subject's during the trial.
Time Frame: 12 weeks
Population: Full set
Measure: Count of Participants; unit: Participants
Arm/Group | Single Dose of PolyPEPI1018 CRC Vaccine | Multiple Dose of PolyPEPI1018 CRC Vaccine
Number analyzed (Participants) | 5 | 6
Participants | 4 | 5

6. Other Pre Specified Outcome: Number of Participants Having Induced Recruitment of TILs
Description: Assessments of TILs was performed using IHC (Immunoscore CR) CD3/CD8 testing on liver biopsy tissue samples obtained from subjects during a time course from baseline until the Last Visit. The CD3+ and CD8+ cell densities were determined in the core tumor and invasive margin using Immunohistochemistry (IHC) staining followed by digital pathology.
Time Frame: Last visit, up to 38 weeks
Population: Only subjects who had tissue-pairs for TIL measurements (4 of 11).
Measure: Count of Participants; unit: Participants
Groups:
- Single Dose of PolyPEPI1018 CRC Vaccine: by sample quality only 2 of 5 single dosed patients were tested for PolyPEPI1018 induced recruitment of TILs (CD3+ and CD8+ T cells) to the invasive margin and core tumor area
- Multiple Dose of PolyPEPI1018 CRC Vaccine: by sample quality only 2 of 6 multiple dosed patients were tested for PolyPEPI1018 induced recruitment of TILs (CD3+ and CD8+ T cells) to the invasive margin and core tumor area
Arm/Group | Single Dose of PolyPEPI1018 CRC Vaccine | Multiple Dose of PolyPEPI1018 CRC Vaccine
Number analyzed (Participants) | 2 | 2
Participants | 1 | 2

ADVERSE EVENTS:
Time Frame: up to 41 weeks
Arm/Group | Single Dose of PolyPEPI1018 CRC Vaccine | Multiple Dose of PolyPEPI1018 CRC Vaccine
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/6
Serious Adverse Events (participants affected / at risk) | 1/5 | 2/6
Other Adverse Events (participants affected / at risk) | 2/5 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Dose of PolyPEPI1018 CRC Vaccine (N=5) | Multiple Dose of PolyPEPI1018 CRC Vaccine (N=6)
THROMBOEMBOLIC EVENT (Embolism) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
ABDOMINAL PAIN (Abdominal pain) (Gastrointestinal disorders) | 0 (0) | 1 (1)
BOWEL OBSTRUCTION (Intestinal obstruction) (Gastrointestinal disorders) | 0 (0) | 1 (1)
NON-INFECTIOUS ACUTE ENCEPHALITIS (Noninfective encephalitis) (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Dose of PolyPEPI1018 CRC Vaccine (N=5) | Multiple Dose of PolyPEPI1018 CRC Vaccine (N=6)
INJECTION SITE REACTION-SOME SUBCUTANEOUS NODULARITY (General disorders) | 1 (1) | 3 (4)
MUSCLE DISORDERS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
NEUROLOGICAL DISRORDERS NEC (Nervous system disorders) | 1 (1) | 0 (0)
ANAEMIAS NONHAEMOLYTIC AND MARROW DEPRESSION (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
GASTROINTESTINAL MOTILITY AND DEFAECATION CONDITIONS (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTROINTESTINAL SIGNS AND SYMPTOMS (Gastrointestinal disorders) | 0 (0) | 1 (1)
JOINT DISORDERS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
EMBOLISM AND THROMBOSIS (Vascular disorders) | 0 (0) | 1 (1)
GENERAL SYSTEM DISORDERS NEC (General disorders) | 0 (0) | 1 (1)
EPIDERMAL AND DERMAL CONDITIONS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
CENTRAL NERVOUS SYSTEM INFECTIONS AND INFLAMMATIONS (Nervous system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-04-10): https://cdn.clinicaltrials.gov/large-docs/32/NCT03391232/Prot_SAP_001.pdf
  • Informed Consent Form (2018-09-07): https://cdn.clinicaltrials.gov/large-docs/32/NCT03391232/ICF_000.pdf